CLINICAL TRIAL: NCT01447797
Title: Single Dose Open-label Comparative Pharmacokinetic Study to Assess the Pharmacokinetic Characteristics of Irbesartan and Atorvastatin Between Irbesartan/Atorvastatin Combination Tablet and Coadministration of Irbesartan and Atorvastatin Tablets in Healthy Male Subjects
Brief Title: A Bioequivalence Study Comparing Irbesartan/Atorvastatin Combination Tablet With Coadministration of Irbesartan and Atorvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-IBAT-104
Record Dates: First submitted 2011-09-28; First posted 2011-10-06 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: Irbesartan; Atorvastatin; combination
MeSH Terms: interventions — Irbesartan; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP0912 (Experimental): Irbesartan/Atorvastatin combination tablet
  Interventions: Drug: HCP0912 / Irbesartan and Atorvastatin
- Irbesartan and Atorvastatin (Active Comparator): coadministration of irbesartan and atorvastatin
  Interventions: Drug: HCP0912 / Irbesartan and Atorvastatin

INTERVENTIONS:
Drug: HCP0912 / Irbesartan and Atorvastatin — Irbesartan and Atorvastatin combination tablet / coadministration of Irbesartan and Atorvastatin

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics and safety after oral administration of Irbesartan and Atorvastatin in combination as HCP0912

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 45
* Signed informed consent form
* weight : over 45kg and in the range of ±20% of IBW

Exclusion Criteria:

* Has a medical history of hypersensitivity to atorvastatin or irbesartan
* severe Hypotension
* Not eligible for subject in health examination within 28 days of IP administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
AUC of Irbesartan | 0-48 hrs
AUC of Atorvastatin and 2-hydroxy atorvastatin | 0-48 hrs
Cmax of Irbesartan | 0-48 hrs
Cmax of Atorvastatin and 2-hydroxy atorvastatin | 0-48 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea